CLINICAL TRIAL: NCT03445754
Title: Effect of Transcutaneous Vagal Stimulation (TVS) on Endothelial Function and Arterial Stiffness in Peripheral Artery Disease
Brief Title: Effect of Transcutaneous Vagal Stimulation (TVS) on Endothelial Function in PAD
Acronym: TVS-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 8473
Record Dates: First submitted 2017-10-12; First posted 2018-02-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease; Endothelial Dysfunction; Autonomic Imbalance
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This is a pilot study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding will be done so the investigator performing the FMD, LSCI and PWA testing will be blinded to the allocation of TVS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional Arm (Experimental): Active TVS will be performed by use of a Tragus stimulator device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour.
  Interventions: Device: TVS
- Control (Sham Comparator): Sham TVS will be performed by use of a Tragus stimulator device with electrodes attached to the ear lobule. Stimulator will be applied continuously for 1 hour.
  Interventions: Device: Sham TVS

INTERVENTIONS:
Device: TVS — Active TVS will be performed by use of a Tragus stimulator device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour
  Arms: Interventional Arm
Device: Sham TVS — Device will be applied but not to the Tragus of the ear but will be attached to the ear lobule.
  Arms: Control

SUMMARY:
Peripheral arterial disease (PAD) constitutes a major public health burden. The incidence of PAD increases with age and is associated with other comorbid cardiovascular disorders. Atherosclerosis which underlies PAD is associated with increased arterial stiffness and an enhanced inflammatory state as evidenced by increased levels of pro-inflammatory cytokines and markers. One the earliest signs of cardiovascular disease is endothelial dysfunction which is characterized by a decreased vasodilatory capacity of the vascular endothelium and this lesion predates the development of clinical atherosclerosis. Endothelial dysfunction has been shown to be widely prevalent in PAD. It is postulated that endothelial dysfunction is due to enhanced sympathetic drive, diminished parasympathetic drive, chronic inflammatory state all of which leads to reduced nitric oxide synthase activity in the vascular endothelium with subsequent loss of vasodilatory capacity. Studies have shown endothelial dysfunction to be reversible with pharmaco-therapeutic interventions, though these interventions are associated with their own adverse effects. Stimulation of Vagal nerve increases the parasympathetic activity while suppressing sympathetic drive, decreases inflammation and enhancing nitric oxide synthase activity. Recent experimental and clinical data suggest that low-level tragus nerve stimulation (by stimulating the auricular branch of the vagus nerve located at the tragus of the external ear) may produce the same desired neuromodulator effect compared to vagus nerve stimulation. It is however unknown if Transcutaneous Vagal Stimulation (TVS) would lead to improved endothelial function as measured by flow mediated dilatation (FMD) and laser speckle contrast imaging(LSCI), a non-invasive method of measuring endothelial function or decrease in arterial stiffness as measured by Pulse Wave Analysis (PWA), in patients with PAD. The objective of this study is to determine the impact of TVS on endothelial dysfunction as measured by FMD & LSCI and arterial stiffness. Study population will include patients with established diagnosis of PAD. After performing baseline FMD, LSCI and PWA patients will be randomized to TVS and sham stimulation with cross over. The patient randomized to TVS stimulation will obtain stimulation for 1 hour followed by measurement of FMD,LSCI and PWA. There will be a washout period of at least 24 hours with patient crossing over to the other arms thus serving as their self-control.

ELIGIBILITY:
Inclusion Criteria:

1. peripheral arterial disease (PAD) - patients with an ankle-brachial index of <0.9
2. symptoms of intermittent claudication, rest pain, or minor tissue loss (Rutherford category I-V)

Exclusion Criteria:

1. patients with acute limb ischemia
2. Patients with overt congestive heart failure / recent acute myocardial infarction (< 3 months)
3. Premenopausal women and post-menopausal women on hormone supplements.
4. chronic inflammatory disease (systemic lupus erythematosus, rheumatoid arthritis, and Crohn's disease), or receiving therapy with steroids, cyclosporine, methotrexate or immunocompromised patients.
5. unilateral or bilateral vagotomy
6. Patients with bilateral upper extremity amputation
7. pregnant patients
8. prisoners
9. end-stage renal disease.
10. End-stage liver disease.
11. patients with BMI>34
12. Patients with upper extremity arterial disease
13. history of recurrent vasovagal syncope, Sick sinus syndrome, 2nd- or 3rd-degree atrioventricular block (AV) block, prolonged first degree AV block.
14. Refusal to sign a consent form.
15. Significant hypotension from autonomic dysfunction
16. Patients with pacemakers who have significant interaction with TVNS during testing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Flow mediated vasodilatation | Change from baseline to post stimulation(within 10 minutes of stimulation) with TVS/Sham stimulation
  Flow mediated vasodilatation will be tested. A change in the maximal diameter of the brachial artery(in mm) will be assessed immediately(within 10 minutes) after TVNS/sham stimulation.

SECONDARY OUTCOMES:
Endothelial function in microcirculation | Change from baseline to post stimulation(within 20-30 minutes of stimulation) with TVS/Sham stimulation
  LSCI based calculation of perfusion unit before and after TVS/Sham stimulation
Pulse wave analysis | Change from baseline to post stimulation(within 15-20 minutes) with TVS/Sham stimulation.
  Arterial elasticity. Augmentation pressure (AP) will be calculated which is expressed as a percentage of the aortic pulse pressure (PP) which is the difference of systolic and diastolic BP(mm Hg).

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Dasari, MD, MPH, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided